CLINICAL TRIAL: NCT07051577
Title: The Effect of Neuroscience-Based Exercise Training on Shooting Performance and Neuromuscular Performance in Archers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Şule Şahin, Principal Investigator (PhD student in Physiotherapy), Istinye University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstinyeUnv2025
Record Dates: First submitted 2025-06-18; First posted 2025-07-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Archery; Physiotherapy and Rehabilitation; Muscle Activity; Visual Rehabilitation; Core Stabilization Exercise Therapy
Keywords: archery; physiotherapy and rehabilitation; Sports Vision Training; balance; core stabilization exercise therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): There are standard exercise programs consisting of scapular stabilization and balance exercises.These exercises are commonly used in clinical rehabilitation and will not include any additional neurosensory or visual components.
  Interventions: Other: control group
- Intervention group (Experimental): Participants will receive neuroscience-based exercise training under researcher supervision, twice a week for 6 weeks. The program includes gaze stabilization, scapular and core stabilization, balance training, and NeuroTracker exercises in three progressive phases.
  Interventions: Other: Exercise Group

INTERVENTIONS:
Other: Exercise Group — Participants in the neuromuscular exercise group will undergo a training program supervised by the researcher, conducted twice a week for 6 weeks. This group will receive gaze stabilization training, core stabilization training, scapular stabilization training, balance training, and NeuroTracker training.
  The exercises provided to the neuromuscular exercise group are structured in three phases and progressively intensified based on phase transition criteria.
  Arms: Intervention group
Other: control group — There are standard exercise programs consisting of scapular stabilization and balance exercises.These exercises are commonly used in clinical rehabilitation and will not include any additional neurosensory or visual components.
  Arms: Control group

SUMMARY:
Archery is a sport that demands sport-specific motor performance, emphasizing fine motor control, postural stability, balance, and concentration skills. Athletes aim to deliver the arrow to the target by ensuring maximum stability with minimal body movement during shooting. While muscle strength, upper extremity endurance, and overall body stability are among the primary factors influencing performance, many other parameters also determine shooting success. Studies investigating muscle activity in archery have demonstrated that the primary muscle groups involved in shooting are the scapular muscles, shoulder girdle muscles, and forearm muscles. These muscles are activated at varying levels to facilitate target focus and play an active role in shooting by contributing to postural and scapular stabilization. Additionally, core muscles enhance movement capacity by centrally stabilizing the body during motion. Activation of pelvic-region muscles, in particular, contributes to improved balance skills, thereby making a meaningful impact on performance.

Archers are expected to maintain stability by minimizing movement during shooting and to rapidly adapt to postural instability that may arise during aiming. Every involuntary movement decreases stability and makes it harder to hit the center of the target. In this context, executing motor actions with high precision and developing adaptive responses to postural instability are of great importance. One of the core components of the balance system-the visual system-also significantly affects performance. During postural sway, visual stabilization plays a critical role; as the distance to the target increases, displacements on the retina become larger, making visual focusing more challenging. Moreover, to make the shooting decision at the right moment, it is essential to maintain visual concentration effectively.

In this project, while no intervention will be applied to the control group, archers using classical bows in the exercise group will participate in a six-week neuroscience-based exercise program. The program includes scapular and core stabilization, balance training, gaze stabilization, and NeuroTracker training. This six-week program is designed to be progressive and holistic, and its effects will be investigated.

Muscle activity will be analyzed through EMG, postural sway will be assessed using the ProKin TecnoBody 252 stabilometric platform, clinical upper extremity balance will be evaluated with the Y Balance Test, eye tracking will be measured using the Pupil headset (Pupil Labs), and spinal stabilization endurance will be assessed through the Biering-Sorensen Test, Lateral Bridge Test, and the Step Test. Shooting performance will be evaluated based on target paper scores. Statistical analyses will be performed using IBM SPSS version 28. Both descriptive and inferential statistical methods will be utilized. Within the scope of descriptive statistics, participants' demographic characteristics and other key variables will be summarized using mean (X̄), standard deviation (SD), frequency (n), and percentage (%). The findings will be evaluated at a significance level of p<0.05.

The study will include a comprehensive analysis using objective measurement methods. In the literature, no previous study has approached neuroscience-based exercise interventions for archers in such a comprehensive and multidimensional manner. This project aims not only to enhance athletic performance but also to prevent shoulder, scapular, and upper extremity injuries that may result from repetitive shooting movements. This research will be one of the first comprehensive studies to address balance, muscle activity, and cognitive performance in archery holistically, offering an original and scientifically valuable contribution to the sports science literature.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 15 and 18 years
* Licensed archer using a classical bow for at least 6 months
* Using a clicker for at least 6 months
* Training at least twice a week

Exclusion Criteria:

* Presence of any symptoms related to the upper or lower extremities
* Any type of surgical intervention in the upper extremity or spine
* Presence of mental or cognitive disorders
* Use of substances that may affect shooting performance, such as painkillers, sedatives, or alcohol

Withdrawal Criteria:

* Reporting an injury or illness during the study
* Experiencing acute muscle spasm
* Choosing to discontinue participation
* Failing to attend exercise training sessions on two consecutive occasions

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Shooting Performance | Change from Shooting Performance at 6 weeks
  Each participant will perform two sets of archery shots on a 40 cm target face at an 18-meter shooting range, with 3 arrows per set. Scoring is based on a concentric ring system, with the center worth 10 points, decreasing outward to 9, 8, 7, and 6 points. The total score will be calculated as the sum of all shot values. The aim is to assess shooting accuracy and performance.
Muscle Activity | Change from Muscle Activity at 6 weeks
  Each participant will perform a total of two sets of archery shots-3 arrows per set-at a FITA 40 cm target from an 18-meter shooting distance. During the shooting, EMG data will be recorded. Surface EMG will be used to measure the activation of the anterior, middle, and posterior parts of the M. Deltoideus; the upper, middle, and lower parts of the M. Trapezius; and the M. Serratus Anterior muscle.
Muscle strength | Change in muscle strength over 6 weeks
  Muscle strength of the anterior, middle, and posterior parts of the M. Deltoideus; the upper, middle, and lower parts of the M. Trapezius; and the M. Serratus Anterior will be assessed using a myometer. During the measurement, the participant will be instructed to resist against maximal resistance applied by the examiner.

SECONDARY OUTCOMES:
Postural Sway Assessment | Change from Postural Sway Assessment at 6 weeks
  Stability and limits of stability will be assessed using the ProKin TecnoBody 252 stabilometric platform. This device will be used to evaluate the overall stability index and limits of stability.
Eye Tracking | Change from Eye Tracking at 6 weeks
  Eye tracking is the process of determining the position of eye movement based on the location of gaze or head position. During the experimental shooting task, participants will wear a wearable eye-tracking device (Pupil headset, Pupil Labs GmbH™, Germany). Using this device, saccadic eye movements and the deviation distance of gaze fixation from the center of the target during arrow release will be monitored. The mean values of the recorded data will be calculated for analysis.
Endurance of extensor spinal stabilizer muscles | Change from Endurance of extensor spinal stabilizer muscles at 6 weeks
  Biering-Sorensen Test:
  This test will be conducted to assess spinal stabilization and the endurance of extensor muscles. For the test, the participant will lie in a prone position with the pelvis and lower extremities supported on a table, while the upper body hangs off the edge in a flexed position. After the legs are stabilized using either manual support or a strap, the participant will be instructed to perform trunk extension with arms crossed over the chest and maintain a horizontal position parallel to the ground. The moment they reach full extension will be considered the starting point, and the duration for which the participant can hold this position will be measured with a stopwatch and recorded in seconds.
Endurance of flexor spinal stabilizer muscles | Change from Endurance of flexor spinal stabilizer muscles at 6 weeks
  Sit-Up Test: This test is used to assess the endurance of the trunk flexor muscles. While lying in a supine position, the participant will bend their knees to 90° and keep their arms crossed over the chest. The upper body will be slightly raised until the head, neck, and scapulae lift off the ground, achieving approximately 60° of trunk flexion. The participant will attempt to maintain this position for as long as possible, and the duration until the posture is no longer maintained will be measured in seconds.
Endurance of oblique spinal stabilizer muscles | Change from Endurance of oblique spinal stabilizer muscles at 6 weeks
  Lateral Bridge Test: The test will be performed on both sides-right and left. Athletes will be positioned in a side-lying posture with the tested-side arm perpendicular to the floor, elbow flexed at 90°, and the forearm resting on the surface. The upper arm will be crossed over the chest, the lower extremities extended, and the top foot placed in front of the bottom foot. Participants will be asked to lift their bodies off the ground, supporting themselves on their forearm and feet, and maintain this position. The duration for which they can hold the position before it breaks will be measured with a stopwatch and recorded in seconds.
Balance Assessment | Change from Balance Assessment at 6 weeks
  Balance will also be assessed using the Upper Extremity Y Balance Test.While in a push-up position with both hands placed shoulder-width apart on the test platform, the participant will be instructed to reach the moveable reach indicator as far as possible in the medial, then superolateral, and finally inferolateral directions.

CONTACTS AND LOCATIONS:
Overall Officials: SULE TOPCU SAHIN, PhD (c), Principal Investigator — Istinye University

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of individual participant data (IPD) is currently under consideration. Factors such as ethical approvals, institutional policies, and data privacy regulations are being reviewed before making a final determination.